CLINICAL TRIAL: NCT00413556
Title: Randomised, Double-Blind, Placebo-Controlled Phase IIIb Study Investigating Changes in Immunological Parameters and Cutaneous Reactivity Induced by a Short Course Immunotherapy With ALK Grass Tablets
Brief Title: Changes in the Immune Response and Skin Reactivity of Grass Pollen Allergic Patients Treated With ALK Grass Tablets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Pilar Rico Nieto - Medical Department, ALK-Abelló S.a.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT-16
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Allergy
Keywords: Rhinitis; Oral tablets; Ig G4; grass pollen; inmunotherapy
MeSH Terms: conditions — Hypersensitivity; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: ALK Grass tablet
- 2 (Placebo Comparator)
  Interventions: Biological: ALK Grass tablet

INTERVENTIONS:
Biological: ALK Grass tablet

SUMMARY:
We plan to determine changes in the immune system during the allergic response to grass pollen allergens. We have chosen a particular element of the immune response, the immunoglobulin G4 (IgG4) as an indicator.

We hypothesize that treatment with Grazax will increase serum levels of Phleum pratense specific IgG4 and IgE, as well as reduce the cutaneous sensitivity of the early (IgE mediated) and late (cell mediated) allergic response.

ELIGIBILITY:
Inclusion Criteria:

* A history of grass pollen allergy
* Positive skin prick test to grass
* Positive specific IgE to grass

Exclusion Criteria:

* Treatment with anti-IgE

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Difference in serum leves of IgG4 | 6 months

SECONDARY OUTCOMES:
Changes in IgE level | 6 months
Changes in cutaneous response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Rico, MD, Study Chair — Medical Director, ALK-Abello, S.A.
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain